CLINICAL TRIAL: NCT04110938
Title: Paediatric Early Rehabilitation/Mobilisation During InTensive Care: An Observational Study
Brief Title: Paediatric Early Rehabilitation/Mobilisation During InTensive Care
Acronym: PERMIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: University of Nottingham (Other); Newcastle University (Other); Northumbria University (Other); University of Cambridge (Other); University of Leeds (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: RG_18-161
Record Dates: First submitted 2019-08-14; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-08

CONDITIONS: ICU; Critical Illness
Keywords: PICU; Paediatric; Early mobilisation; Early rehabilitation; Observational
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the UK, critical illness or injury affects about 19,000 Children and Young Persons (CYP) every year who are admitted to the paediatric intensive care unit (PICU) to receive life-sustaining treatments. Although survival rates from PICU are at an all-time high (>96%), low levels of mortality have been offset by an increase in morbidity. The impact of being critically ill and exposed to the PICU is multiple. Weakness, cognitive impairment, organ dysfunction, and psychological problems have been reported to emanate from deconditioning. Subsequently, post-PICU many CYP experience significant and residual physical, cognitive, and psychosocial morbidities that impact on their quality of life. The contemporary focus has turned to the development, testing, and implementation of interventions to minimize the harmful effects of critical care and maximize patient outcomes.

Early rehabilitation and/or mobilisation (ERM) encompasses patient-tailored interventions, delivered individually or in a bundled package, provided by health professionals from multiple disciplines and care-givers within intensive care settings to promote recovery, both physical (e.g. movement, functional activities, ambulation) and non-physical (e.g. speech, play, psychological, cognitive).

Rehabilitation has been shown to improve quality of life and patient outcomes; reduce health inequalities, and make significant savings to the health care system. Benefits have been demonstrated in the use of ERM in adult ICU populations in relation to patient outcomes as well as healthcare utilization. Studies also indicate that the intervention is safe and feasible, reduces delirium and increases ventilator-free days, improves day-to-day functioning and reduces hospital readmissions. However, in the United Kingdom (UK), the understanding of current ERM practices (including content, barriers, facilitators, feasibility, and safety) and their impact on the outcomes of pediatric ICU patients is limited. This has stifled an evidence-based approach to ERM which has resulted in disparity in the adoption and utilization of ERM interventions in PICUs across the UK.

To address this critical gap, the first phase of a four-phase program of the PERMIT study will generate evidence of current PICU ERM practices by conducting a survey and an observational study.

The second phase of the study will involve conducting qualitative workshops to develop a prototype ERM program. Qualitative workshops will also be conducted among key stakeholders (clinicians, parents, CYP) to inform the design of an ERM intervention.

The third phase will investigate this ERM program in a pilot study in UK PICUs and finally, the efficacy of the intervention will be tested using a large scale, definitive randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The PERMIT study aims to ascertain current ERM practices within PICU settings and barriers/facilitators to ERM delivery.

The investigators plan to directly observe current ERM practices within UK PICUs, identify patients who do and do not receive ERM, describe the variation between PICUs and factors associated with ERM practices.

Inclusion Criteria:

1. All Children and Young Persons (CYP) (0-<16 years)
2. Admitted to PICU
3. Remain within PICU on day 3 post-admission

The broad inclusion criteria will allow for the observation of all types of patients admitted for PICU care (acute and elective e.g. post-surgical recovery) and all age ranges.

Exclusion criteria:

1. A local decision by a Principal investigator (PI) or treating clinical team not to include patient
2. Parent or guardian chooses to opt-out

Prospective data about all children admitted to PICU for 3 days or more will be collected. Eligible patients will be identified, screened and enrolled in the study. Posters and patient information leaflets will be provided to parents/legal guardians within participating PICU explaining their rights to withdraw from the study without affecting the future care of their child. Data collected as part of the study will be stored for ten years, in line with Good Clinical Practice (GCP) guidelines. No identifiable data will be collected or shared with the PERMIT study team at any time.

Following the observation of current ERM delivery and identification of patients who may benefit from ERM in selected PICUs, the study investigators will use this information to model how many patients may be available in the UK for a potential future RCT. This will be achieved by modeling patient demographic information with the Paediatric Intensive Care Audit Network (PICANet) dataset.

ELIGIBILITY:
Inclusion Criteria:

* All Children and Young Persons (CYP) (0-<16 years)
* Admitted to PICU
* Remain within PICU on day 3 post-admission

Exclusion Criteria:

* Local decision by PI or treating clinical team not to include patient
* Parent or guardian choose to opt out.

Ages: 38 Weeks to 16 Years | Sex: All
Age Groups: Child
Study Population: All Children and Young Persons (CYP) (0-<16 years) admitted to paediatric itnesive care units for 3 days or more
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-28 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of early rehabilitation and/or mobilisation (ERM) delivered on Day 3 post PICU admission | 3 weeks
  The prevalence and scope of ERM will be described as the proportion of patients with any 'active interaction' delivered on Day 3 post-admission.

SECONDARY OUTCOMES:
Incidence rates and ratios of the number of ERM interventions from Day 3 to Day 10 post PICU admission | 3 weeks
  Incidence rates will be calculated and exploratory analysis will be performed to understand factors associated with the incidence of ERM delivery.
The cumulative prevalence of ERM for each day in PICU after Day 3 up to Day 10 post-admission | 3 weeks
  The cumulative prevalence for each day in PICU after Day 3 up to Day 10 post-admission with whom ERM may/may not be appropriate will be calculated.
  Exploratory analysis will be performed to understand factors associated with the incidence of ERM delivery.
Factors associated with variability of early rehabilitation and/or mobilisation (ERM) delivery | 3 weeks
  Exploratory analysis will be performed to understand factors associated with ERM delivery. ERM delivered per patient will be quantified as well as the characteristics of patients receiving ERM, type of ERM interventions delivered and factors associated with variability of delivery between PICUs will be explored.
To evaluate predictors of ERM provided on Day 3 post-PICU-admission | 3 weeks
  Exploratory analysis will be used to explore the characteristics of patients receiving ERM on Day 3 post-PICU-admission.
  Multilevel multivariable regression models will be used to evaluate predictors of ERM provision
Dose of ERM per day of PICU admission | 3 weeks
  Exploratory analysis will be performed to quantify the dose (duration, measured in minutes) of ERM for each day over the 3-week period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby Scholefield, Dr, Study Chair — Birmingham Women's and Children's Hospital
Locations (1):
- Birmingham Women's and Children's Hospital PICU, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Scholefield BR, Menzies JC, McAnuff J, Thompson JY, Manning JC, Feltbower RG, Geary M, Lockley S, Morris KP, Moore D, Pathan N, Kirkham F, Forsyth R, Rapley T. Implementing early rehabilitation and mobilisation for children in UK paediatric intensive care units: the PERMIT feasibility study. Health Technol Assess. 2023 Nov;27(27):1-155. doi: 10.3310/HYRW5688. PMID 38063184